CLINICAL TRIAL: NCT03004677
Title: Effect of Skin-to-skin Contact on Interaction and Parents' Sleep
Acronym: Neo-SIPaS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To difficult to recruit.
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Evalotte Morelius, Associate professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Linkoeping University
Record Dates: First submitted 2016-12-10; First posted 2016-12-29 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Sleep Quality; Communication; Stress Reaction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Communication; Fractures, Stress | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous skin-to-skin contact (Experimental): Infants assigned to SSC will rest skin-to-skin on parents' chest 24 hours a day for four days alternating between the parents.
  Interventions: Behavioral: Continuous skin-to-skin contact
- Standard Care (Active Comparator): Infants and parents will receive standard care provided in the NICU
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Continuous skin-to-skin contact — Infants will rest in skin-to-skin contact on parents' chest 24 hours a day alternating between the parents. The parents will note who provides the SSC and if and for how long they are off SSC for any reason.
  Arms: Continuous skin-to-skin contact
Other: Standard Care — Infants will receive regular care in the NICU. Parents may practice SSC if they like. Parents will note if, with whom, and for how long they provide SSC.
  Arms: Standard Care

SUMMARY:
This study evaluates the effect of a late intervention of continuous skin-to-skin contact (SSC) in the neonatal intensive care unit (NICU). Half of the participants will receive the intervention and the other half will receive standard care.

DETAILED DESCRIPTION:
The intervention is based on a method developed to facilitate closeness and human touch between parents and preterm infants in neonatal intensive care. Continuous skin-to-skin contact (SSC) means, in this study, that the late preterm infant is cared for skin-to-skin on the parents' chest, instead of in a heating-bed, 24 hours a day. The parents will take turns to care for the infant in SSC.

ELIGIBILITY:
Inclusion Criteria:

* Parents staying at the NICU with a single preterm infant born <33 weeks of gestation
* The family should have been transferred to family-room from intensive care
* Swedish speaking parents

Exclusion Criteria:

* Infants with major congenital malformation,
* Infants with intraventricular hemorrhage grade III-IV
* Infants with chromosome defect that could affect the infant´s ability to interact.
* Parents with sleeping disorder
* Parents with psychiatric problem or drug use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Day 1 to 5
  sleep diary every day for five days

SECONDARY OUTCOMES:
Mood | day 2 to 5
  Mood Adjective Checklist (MACL)
Bonding | Baseline and 1-3 days before planned discharge from the NICU.
  Mother to Infant Bonding Scale (MIBS)
Depression | Baseline and 1-3 days before planned discharge from the NICU.
  The Edinburgh Postnatal Depression Scale, EPDS
Anxiety | Baseline and 1-3 days before planned discharge from the NICU.
  State Trait Anxiety Inventory, STAI
Activity | Day 1-5
  Actigraph every day for five days

CONTACTS AND LOCATIONS:
Overall Officials: Evalotte Mörelius, PhD, Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - University Hospital, Linköping
  - University hospital Örebro, Örebro
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morelius E, Olsson E, Sahlen Helmer C, Thernstrom Blomqvist Y, Angelhoff C. External barriers for including parents of preterm infants in a randomised clinical trial in the neonatal intensive care unit in Sweden: a descriptive study. BMJ Open. 2020 Dec 4;10(12):e040991. doi: 10.1136/bmjopen-2020-040991. PMID 33277288
- [Derived] Angelhoff C, Blomqvist YT, Sahlen Helmer C, Olsson E, Shorey S, Frostell A, Morelius E. Effect of skin-to-skin contact on parents' sleep quality, mood, parent-infant interaction and cortisol concentrations in neonatal care units: study protocol of a randomised controlled trial. BMJ Open. 2018 Aug 1;8(7):e021606. doi: 10.1136/bmjopen-2018-021606. PMID 30068615